CLINICAL TRIAL: NCT07035717
Title: How do Adults Sexual Offender Against Pre-pubescent Minors Perceive the Notion of Consent Based on the Account of Their Lived Experience ?
Brief Title: How do Adults Sexual Offender Against Pre-pubescent Minors Perceive the Notion of Consent Based on the Account of Their Lived Experience ? (SOconsent)
Acronym: SOconsent
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL25_0222
Record Dates: First submitted 2025-05-28; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Violence Against Children; Sexual Violence; Consent
Keywords: forensic psychiatry; sexual violence against minors; consent; prevention of sexual violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRIAVS-LR patient: Purposeful sampling of adult perpetrators of sexual offenses against prepubescent minors, followed at the CRIAVS-LR (Resource Center for Professionals Working with Perpetrators of Sexual Violence in Languedoc-Roussillon)
  Interventions: Other: Patient interview

INTERVENTIONS:
Other: Patient interview — A semi-structured interview with five questions will be conducted, with audio recording, which will later be transcribed verbatim.

SUMMARY:
In 2024, the police and gendarmerie recorded 12,260 victims of sexual violence, an increase of 7% compared with 2023. In 2019, 36,000 cases of sexual violence (rape or sexual assault) were handled by the public prosecutor's office. In 53.3% of cases, sexual violence was committed against minors. In 95% of cases, the perpetrators were male. The word is getting out about sexual violence, bringing the subject of consent to the forefront of media and scientific news. Even if the word is common, its definition is subtle, its understanding complex and many factors can influence its perception, including sex education, psychosocial skills and adherence to gender stereotypes.

Research has shown that most people define sexual consent in the context of an oral conversation. However, studies show us that this is not what is done in practice: sexual consent or refusal is most often non-verbal and indirect.

No studies have been carried out on consent in a population of perpetrators of sexual violence against minors.

It is know that perpetrators of sexual violences exhibit alexythmias and cognitive distortions in the area of sexuality. The issue of consent is crucial, since perpetrators of sexual violences may believe that prepubescent children are capable of consenting to a sexual act.

The aim of this study is to obtain a better analysis of the mechanisms, situations, facilitating factors, representations, sensitive perceptions and attitudes that lead perpetrators of sexual violences of minors to experiment with consent in their relationships. A better assessment of their understanding of consent and the factors that may have influenced it could have an impact on primary, secondary and tertiary prevention, as well as on treatment, and avoid potential new acts.

ELIGIBILITY:
Inclusion Criteria:

* adult perpetrators of sexual offences against prepubescent minors followed up at CRIAVS-LR

Exclusion Criteria:

* Subjects with dementia, intellectual disability or decompensated psychiatric disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rational sampling of adult perpetrators of sexual offences against prepubescent minors followed up at the CRIAVS-LR (Resource Centre for Interveners with Perpetrators of Sexual Violence in Languedoc Roussillon)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
One guided interview to measure the consent perception of patient | Baseline single time point
  The objective of this study is to understand the determinants of consent perception among individuals who have committed sexual violence against minors, based on the collection of their lived experiences. The interviews will be analyzed using a phenomenological approach, aiming to generate data from the lived experiences captured in the verbatim transcripts, in order to identify categories related to the phenomenon under study-namely, consent-each representing a distinct dimension of it. This analysis will be structured in several stages. Raw data will be compiled in a Word document.
  Following segmentation into meaning units and thematization through an inductive coding process and classificatory logic, the analysis will focus on identifying elements relevant to the research question, with particular attention to predefined indicators (such as empathy, coercion, cognitive distortions, and negative past experiences related to consent).

SECONDARY OUTCOMES:
Socio-demographic data | Baseline single time point
  age (year), criminal records, marital status, study level

CONTACTS AND LOCATIONS:
Overall Officials: Céline BAIS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UH MONTPELLIER - La Colombiere CRIAVS, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided